CLINICAL TRIAL: NCT00924274
Title: Effect of a Diet With Rapeseed Oil /Sunflower Oil on Lipoprotein in Children and Adolescents With Familial Hypercholesterolemia
Brief Title: Effect of Rapeseed Oil and Sunflower Oil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Kurt Widhalm/Prof., Devision Nutrition and Metabolsim, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EROSO
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Rapeseed Oil; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental)
  Interventions: Dietary Supplement: rapeseed oil
- sunflower oil (Active Comparator)
  Interventions: Dietary Supplement: sunflower oil

INTERVENTIONS:
Dietary Supplement: rapeseed oil — rapeseed oil in amounts between 14 and 27 g
  Arms: Lifestyle counseling
Dietary Supplement: sunflower oil — sunflower oil
  Arms: sunflower oil

SUMMARY:
Familial hypercholesterolemia (FH), an inherited disorder of lipoprotein metabolism, is a risk for early cardiovascular disease (CVD). This autosomal dominant disease is characterized by markedly elevated plasma concentrations of low density lipoprotein (LDL) and total cholesterol (TC). The purpose of this study is to compare the effect of a diet low in saturated fats but enriched either with rapeseed oil (RO) or sunflower oil (SO) in children and adolescents with FH on serum lipoproteins.

ELIGIBILITY:
Inclusion Criteria:

* chilren and adolescents between 6 and 18 years of age
* LDLc > 130 mg/dl and
* TC > 200 mg/dl
* 7 day nutrition record
* written informed consent

Exclusion Criteria:

* overweight
* underweight
* mental disability
* drug therapy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Blood analysis including fasting serum lipoproteins (TC, LDLc; HDLc; TG, Lp(a), Apolipoprotein A-1, Apolipoprotein B, BB, hs-CRP, GOT, GPT, GGT, acid composition of plasma lipids. | done in Week 1, Week 7, Week 13

SECONDARY OUTCOMES:
Motivation, compliance, increase of quality of life. | done in Week 1 and Week 13
Acceptance and approach to the disease. | done in Week 1 and Week 13
Improvement of knowledge and understanding about the disease by the patients. | done in Week 1 and Week 13

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Nutrition and Metabolism, Department of Pediatrics, Medical University of Vienna, Vienna, Vienna, Austria